CLINICAL TRIAL: NCT07187856
Title: A Phase 2 Randomised Controlled Study to Investigate the Efficacy and Safety of Subcutaneously Administered PG-102 for 24 Weeks Compared With Placebo and Open-Label Semaglutide in Patients With Type 2 Diabetes Mellitus
Brief Title: Phase 2 Randomized Study of PG-102 vs Placebo and Semaglutide in Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ProGen. Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG-102-P2-WW-01
Record Dates: First submitted 2025-08-28; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: PG-102 and Placebo are administered double-blind; the Semaglutide comparator arm is open-label.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PG-102 (Experimental): Participants receive PG-102 administered subcutaneously once weekly with dose titration.
  Interventions: Drug: PG-102
- Placebo (Placebo Comparator): Participants receive matching placebo administered subcutaneously once weekly.
  Interventions: Drug: Placebo
- Semaglutide (Active Comparator): Participants receive open-label semaglutide administered subcutaneously once weekly, titrated to 1.0 mg.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: PG-102 — PG-102 is administered subcutaneously once weekly with a titration regimen.
  Arms: PG-102
Drug: Placebo — Placebo is administered subcutaneously once weekly.
  Arms: Placebo
Drug: Semaglutide — Open-label semaglutide is administered subcutaneously once weekly with titration regimen.
  Arms: Semaglutide

SUMMARY:
Phase 2 Randomized Study of PG-102 vs Placebo and Semaglutide in Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent before any study-related activities are performed and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
* Adult males and females, 18 to 75 years of age (inclusive) on the day of signing the informed consent form (ICF).
* Must have a diagnosis of T2DM for at least 6 months before screening based on the disease diagnostic criteria.
* Must have an HbA1c value at screening of ≥7.0% and ≤10.0% (≥53 and ≤86 mmol/mol) and treated with diet and exercise alone or a stable dose of metformin (either immediate release or extended release, ≥1000 mg/day and not more than the locally approved dose) for at least 3 months prior to screening.
* Body mass index (BMI) ≥25 to <40 kg/m2 at screening.

Exclusion Criteria:

* Have a diagnosis of type 1 diabetes.
* History of severe hypoglycaemia and/or hypoglycaemia unawareness within 6 months prior to screening.
* Have active proliferative diabetic retinopathy or history of uncontrolled and potentially unstable diabetic retinopathy or maculopathy.
* History of or current chronic pancreatitis, or acute pancreatitis within the past 6 months prior to screening.
* Diagnosis of gastroparesis or history of bariatric surgery or a clinically significant gastric emptying abnormality, in the opinion of the investigator (or delegate).
* Have known liver disease or obvious clinical signs or symptoms of liver disease, including acute or chronic hepatitis; or have any of the following at screening: ALT ≥ 3 × ULN, AST ≥ 3 × ULN, and total bilirubin ≥2 × ULN.
* Concomitant therapy in addition to metformin therapy with another oral antihyperglycaemic medication (OAM) including, but not limited to, sulfonylureas, dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose cotransport 2 inhibitors, alpha-glucosidase inhibitors, and meglitinides. Participants may be randomised if the additional OAM was discontinued at least 3 months prior to screening.
* Have used insulin for diabetic control within the prior year; however, short-term use of insulin for acute conditions is allowed (≤14 days) in certain situations, such as during a hospitalisation or perioperatively.
* Have had any exposure to GLP-1 analogues (including combination products) or other related compounds within the prior 3 months prior to screening, or any history ever of allergies to these medications. Patients who previously took GLP-1 analogues or related compounds and who discontinued those medications for intolerability or lack of efficacy will not be randomised.
* Have been treated with prescription drugs that promote weight loss or similar body weight loss medications including over-the-counter medications within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Absolute change in HbA1c From Baseline at Week 24 | 24 weeks
  Mean absolute change in glycated hemoglobin (HbA1c) from baseline to Week 24, comparing PG-102 with placebo.

SECONDARY OUTCOMES:
Absolute change in HbA1c from baseline to 12 weeks | 12 weeks
  Mean absolute change in HbA1c from baseline to Week 12.
Absolute Change in Body Weight From Baseline at Week 12 and 24 | 12 and 24 weeks
  Mean absolute change in body weight from baseline to Weeks 12 and 24.
Percent Change in Body Weight From Baseline at Week 12 and 24 | 12 and 24 weeks
  Mean percent change in Body Weight from baseline to Week 12 and 24.
Change in Fasting Plasma Glucose (FPG) From Baseline at Week 12 and 24. | 12 and 24 weeks
  Mean change in fasting plasma glucose (mg/dL) from baseline to Week 12 and 24.
Change in 7-Point Self-Monitored Plasma Glucose (SMPG) Profile at Week 12 and 24. | 12 and 24 weeks
  Mean change in the 7-point SMPG profile from baseline to Week 12 and 24.
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 24 weeks
  Number and percentage of participants experiencing TEAEs, SAEs, and discontinuations due to adverse events.
Incidence of Adverse Events of Special Interest (AESIs) - Gastrointestinal | 24 weeks
  Incidence and severity of GI-related AESIs (e.g., nausea, vomiting, diarrhea).
Incidence of anti-drug antibodies (ADA) to PG-102 | 24 weeks
  Number and percentage of participants developing anti-drug antibodies against PG-102.

CONTACTS AND LOCATIONS:
Locations (1):
- Emeritus Research, Camberwell, Victoria, Australia